CLINICAL TRIAL: NCT01148732
Title: Tracheal Rapid Ultrasound Exam (T.R.U.E) for Confirming Endotracheal Tube Placement in Emergency Intubation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Wan-Ching Lien/M.D., National Taiwan University Hospital
Other Study IDs: 201003027R
Record Dates: First submitted 2010-06-08; First posted 2010-06-22 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Intubation
Keywords: Endotracheal tube; ultrasonography
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient needed intubation in emergency department
  Interventions: Procedure: ultrasonography

INTERVENTIONS:
Procedure: ultrasonography — a Toshiba 3.75 MHz convex ultrasonography transducer (Toshiba SSA-550A, Tochigi-ken, Japan) was placed transversely on the anterior neck just superior to the suprasternal notch and bilateral hemithorax by one of two emergency physician during emergency intubation investigators.

SUMMARY:
Reliable endotracheal tube (ETT) insertion confirmation is essential for critically ill patients. Incorrect placement causes a high rate of mortality and morbidity. Therefore, early detection of accidental esophageal intubation must be a primary focus of emergency airway efforts in emergency department (ED). Although many techniques have been suggested to verify the ETT placement, there is currently no entirely reliable method. Ultrasonography (US) is an indispensable and easily accessible tool in ED. Several studies of ultrasonographic confirmation of ETT position provided promising results in cadaver model or patient in a controlled operating room setting.In this study, the investigators have proposed a protocol called T.R.U.E, an acronym for tracheal rapid ultrasound exam, to confirm the ETT position in emergency intubation. This method provided a fast, real-time examination to prevent esophageal or endotracheal intubation.

DETAILED DESCRIPTION:
Establishing a definite airway, endotracheal tube placement, is an important component for resuscitation. A high rate of morbidity and mortality was reported for unrecognized esophageal intubation. Therefore, early detection of esophageal intubation is essential for emergency airway management. There are several methods being used for endotracheal tube confirmation, such as auscultation of breathing sound, chest X-ray and capnography.2 However, all of these methods had false-negative rates and not entirely reliable during resuscitation. Ultrasound is an indispensable and easily accessible tool in emergency department. Recent studies showed that ultrasound can be used to confirm endotracheal tube placement in cadaver model. In this prospective study, we investigate the sensitivity and specificity of ultrasound for endotracheal tube confirmation in emergency intubation The study is conducted in the emergency department at National Taiwan University Hospital and approved by the hospital institutional review board. During resuscitation, the duty emergency resuscitation team performs the intubation and confirms the endotracheal tube position by auscultation and end-tidal capnography. Meanwhile, the researcher performs ultrasonography examinations for endotracheal tube position. A curvilinear ultrasonography transducer is used and placed transversely on the anterior neck just superior to the suprasternal notch and bilateral hemithorax. The result of ultrasonography will be compared with auscultation, capnography and chest X-ray. Sensitivity and specificity of ultrasonography examination is computed to determine the accuracy and effectiveness of clinical use.

ELIGIBILITY:
Inclusion Criteria:

* Patients required intubation

Exclusion Criteria:

* Head and Neck trauma
* Head and Neck tumor
* Status post tracheostomy
* Status post neck surgery
* Children (<18 years old)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient needed emergency intubation in emergency department
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
The endotracheal tube position | 5 minutes
  We use ultrasound to confirm the endotracheal tube position in emergency intubation

SECONDARY OUTCOMES:
Time required for each assessment | 1 hour
  Time required for ultrasonoraphy, capnography and chest X-ray

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Ching Lien, M.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chou HC, Tseng WP, Wang CH, Ma MH, Wang HP, Huang PC, Sim SS, Liao YC, Chen SY, Hsu CY, Yen ZS, Chang WT, Huang CH, Lien WC, Chen SC. Tracheal rapid ultrasound exam (T.R.U.E.) for confirming endotracheal tube placement during emergency intubation. Resuscitation. 2011 Oct;82(10):1279-84. doi: 10.1016/j.resuscitation.2011.05.016. Epub 2011 Jun 1. PMID 21684668